CLINICAL TRIAL: NCT06049173
Title: Evaluation of the Effect of Novel Recruitment Maneuver Therapy for Postoperative Pulmonary Atelectasis in the Patients With Cardiac Surgery
Brief Title: Evaluation of the Effect of Novel Recruitment Maneuver Therapy for Postoperative Pulmonary Atelectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jilai Xiao (Other)
Responsible Party: Sponsor-Investigator, Jilai Xiao, associate chief physician, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: KY20230829-04
Record Dates: First submitted 2023-09-10; First posted 2023-09-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pulmonary Atelectasis; Negative Pressure Therapy
Keywords: Negative extra-abdominal pressure (NEXAP); lung recruitment maneuver; postoperative atelectasis; cardiac surgery
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEXAP group (Experimental): The ventilator mode was changed from SIMV to PSV before LRM. After that, the abdominal pressure cardiopulmonary resuscitation (CPR-LW100) instrument was adopted and adsorbed on the epigastrium of patients. The LRM was performed by pulling up (tension of 20-30 kg) and compressing downward (tension<10 kg) alternately on the abdomen of the patients with a frequency of 12 times per minute to support and maintain breathing. The whole LRM procedure lasted for 3 minutes in total . After LRM, the ventilator mode was changed to its baseline settings.
  Interventions: Device: Negative extra-abdominal pressure (NEXAP)-based lung recruitment maneuver
- PEEP group (Active Comparator): The ventilator mode was changed from SIMV to PSV before LRM. After that, PEEP was increased gradually (every 3-5cmH2O per 30s) from baseline (5-8 cmH2O) to 20cmH2O. The PEEP level was maintained at 20cmH2O for 60s, followed by decrements to baseline PEEP (every 3-5cmH2O per 30s). After LRM, the ventilator was changed to the baseline settings.
  Interventions: Other: stepwise positive end-expiratory pressure (PEEP)-based lung recruitment maneuver

INTERVENTIONS:
Device: Negative extra-abdominal pressure (NEXAP)-based lung recruitment maneuver — The ventilator mode was changed from SIMV to PSV before LRM. After that, the abdominal pressure cardiopulmonary resuscitation (CPR-LW100) instrument was adopted and adsorbed on the epigastrium of patients. The LRM was performed by pulling up (tension of 20-30 kg) and compressing downward (tension<10 kg) alternately on the abdomen of the patients with a frequency of 12 times per minute to support and maintain breathing. The whole LRM procedure lasted for 3 minutes in total. After LRM, the ventilator mode was changed to its baseline settings.
  Arms: NEXAP group
Other: stepwise positive end-expiratory pressure (PEEP)-based lung recruitment maneuver — The ventilator mode was changed from SIMV to PSV before LRM. After that, PEEP was increased gradually (every 3-5cmH2O per 30s) from baseline (5-8 cmH2O) to 20cmH2O. The PEEP level was maintained at 20cmH2O for 60s, followed by decrements to baseline PEEP (every 3-5cmH2O per 30s). After LRM, the ventilator was changed to the baseline settings.
  Arms: PEEP group

SUMMARY:
1. Oxygenation index and bedside ultrasound would be used to evaluate the therapeutic effect of novel recruitment maneuver therapy in the patients with pulmonary atelectasis after cardiac surgery.
2. To establish a new therapy strategy for pulmonary atelectasis after cardiac surgery and to evaluate its effectiveness and safety for the cardiac patients complicated with postoperative pulmonary atelectasis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Underwent cardiac surgery with CPB
* Patients with lung ultrasound evidence of atelectasis after surgery
* Agree to participate in this study by themselves or their family member.

Exclusion Criteria:

* Vasoactive-inotropic score (VIS)>20
* Patients who were not suitable for using abdominal CPR compression-decompression instrument: bleeding from abdominal organs, abdominal aortic aneurysm, large abdominal tumor, intra-abdominal hypertension, etc
* Hemothorax or large pleural effusion confirmed by ultrasonography/X-ray
* Pneumothorax or air leak confirmed by ultrasonography/X-ray
* Considered by other researchers to be unsuitable for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Lung ultrasound score (LUSS) | 5 min before treatment and 5 min after treatment
  The thorax was divided by the anterior axillary line, the posterior axillary line, and a horizontal line beneath the nipple. The intercostal spaces of each of the 12 areas were scanned and analyzed . Aeration loss was assessed by calculating the modified lung ultrasound score (LUSS), which showed sufficient sensitivity to detect aeration loss. Two lung ultrasound examiners provided scores for each area after simultaneous examination of the lung scan. LUSS was then calculated globally (LUSStot， as the sum of the 12 regions score, ranging from 0 to 36), and regionally (LUSSp, posterior, LUSSa, anterior and LUSSl, lateral regions).

CONTACTS AND LOCATIONS:
Overall Officials: Jilai Xiao, Study Director — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ubben JF, Lance MD, Buhre WF, Schreiber JU. Clinical strategies to prevent pulmonary complications in cardiac surgery: an overview. J Cardiothorac Vasc Anesth. 2015 Apr;29(2):481-90. doi: 10.1053/j.jvca.2014.09.020. Epub 2015 Jan 17. No abstract available. PMID 25604600
- [Background] Keogh C, Saavedra F, Dubo S, Aqueveque P, Ortega P, Gomez B, Germany E, Pinto D, Osorio R, Pastene F, Poulton A, Jarvis J, Andrews B, FitzGerald JJ. Non-invasive phrenic nerve stimulation to avoid ventilator-induced diaphragm dysfunction in critical care. Artif Organs. 2022 Oct;46(10):1988-1997. doi: 10.1111/aor.14244. Epub 2022 Apr 12. PMID 35377472
- [Background] Bruni A, Garofalo E, Pasin L, Serraino GF, Cammarota G, Longhini F, Landoni G, Lembo R, Mastroroberto P, Navalesi P; MaGIC (Magna Graecia Intensive care and Cardiac surgery) Group. Diaphragmatic Dysfunction After Elective Cardiac Surgery: A Prospective Observational Study. J Cardiothorac Vasc Anesth. 2020 Dec;34(12):3336-3344. doi: 10.1053/j.jvca.2020.06.038. Epub 2020 Jun 17. PMID 32653270
- [Background] Gattinoni L, Tonetti T, Quintel M. Intensive care medicine in 2050: ventilator-induced lung injury. Intensive Care Med. 2018 Jan;44(1):76-78. doi: 10.1007/s00134-017-4770-8. Epub 2017 Mar 22. No abstract available. PMID 28331959
- [Background] Nielsen J, Ostergaard M, Kjaergaard J, Tingleff J, Berthelsen PG, Nygard E, Larsson A. Lung recruitment maneuver depresses central hemodynamics in patients following cardiac surgery. Intensive Care Med. 2005 Sep;31(9):1189-94. doi: 10.1007/s00134-005-2732-z. Epub 2005 Aug 12. PMID 16096751
- [Background] Scharffenberg M, Wittenstein J, Herzog M, Tauer S, Vivona L, Theilen R, Bluth T, Kiss T, Koch T, Fiorentino G, de Abreu MG, Huhle R. Continuous external negative pressure improves oxygenation and respiratory mechanics in Experimental Lung Injury in Pigs - A pilot proof-of-concept trial. Intensive Care Med Exp. 2020 Dec 18;8(Suppl 1):49. doi: 10.1186/s40635-020-00315-1. PMID 33336263
- [Background] Yoshida T, Engelberts D, Otulakowski G, Katira B, Ferguson ND, Brochard L, Amato MBP, Kavanagh BP. Continuous negative abdominal pressure: mechanism of action and comparison with prone position. J Appl Physiol (1985). 2018 Jul 1;125(1):107-116. doi: 10.1152/japplphysiol.01125.2017. Epub 2018 Mar 29. PMID 29596015
- [Background] Rohrs EC, Bassi TG, Fernandez KC, Ornowska M, Nicholas M, Wittmann JC, Reynolds SC. Diaphragm neurostimulation during mechanical ventilation reduces atelectasis and transpulmonary plateau pressure, preserving lung homogeneity and P ⁢ a O ⁢ 2 / F ⁢ I O 2 . J Appl Physiol (1985). 2021 Jul 1;131(1):290-301. doi: 10.1152/japplphysiol.00119.2021. Epub 2021 Jun 10. PMID 34110233